CLINICAL TRIAL: NCT03907215
Title: A Single-center, Single-blind, Randomized, Placebo-controlled, Sequential Design Phase 1 Study With the Inclusion of Two Double-blind Nested Crossover Parts to Investigate the Drug-drug Interactions Between ACT-541468 and Citalopram in Healthy Male and Female Subjects
Brief Title: A Clinical Study to Examine the Drug-drug Interactions Between ACT-541468 and Citalopram in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: ID-078-114
Record Dates: First submitted 2019-03-21; First posted 2019-04-08 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — daridorexant; Citalopram

STUDY DESIGN:
Intervention Model Description: Single-center, single-blind, randomized, placebo-controlled, sequential design Phase 1 study with the inclusion of two double-blind nested crossover parts
Who Masked: Participant, Investigator
Masking Description: Double-blind to the administration of ACT-541468 (participant). Single- and double-blind to the administration of ACT-541468 (Investigator, single-/double blind is dependent on treatment arm team). Single-blind study with the inclusion of two double-blind nested crossover parts, i.e., subjects will remain blinded to all administrations of ACT-541468.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A and B (Other): On Day 1 and Day 2, subjects will EITHER receive:
  * a single dose of 50 mg ACT-541468 (Treatment A) on Day 1 and a single dose of ACT- 541468 placebo (Treatment B) on Day 2 OR
  * a single dose of ACT-541468 placebo (Treatment B) on Day 1 and a single dose of 50 mg ACT-541468 (Treatment A) on Day 2.
  Interventions: Drug: ACT541468; Drug: ACT541468 placebo
- Treatment C, D, E, and F (Other): From Day 3 to Day 10, subjects will on each day receive:
  • a single dose of 20 mg citalopram and EITHER a single dose of ACT-541468 placebo OR a single dose of 50 mg ACT-541468.
  Interventions: Drug: ACT541468; Drug: ACT541468 placebo; Drug: Citalopram

INTERVENTIONS:
Drug: ACT541468 — 50 mg; film-coated tablet for oral use
Drug: ACT541468 placebo — film-coated tablet for oral use
Drug: Citalopram — 20 mg; tablet tor oral use; for single- or repeated dosing
  Arms: Treatment C, D, E, and F

SUMMARY:
A clinical study to examine the drug-drug interactions between ACT-541468 and citalopram in healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Healthy male and female subjects aged between 24 and 55 years (inclusive) at Screening.
* Body mass index of 18.5 to 29.9 kg/m2 (inclusive) at Screening.
* Women of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1. They must consistently and correctly use a highly effective method of contraception, be sexually inactive, or have a vasectomized partner.
* Women of non-childbearing potential (i.e., postmenopausal, with previous bilateral salpingectomy, bilateral salpingo oophorectomy or hysterectomy, or with premature ovarian failure, XY genotype, Turner syndrome, uterine agenesis).
* Healthy on the basis of physical examination, cardiovascular assessments, and clinical laboratory tests.

Exclusion Criteria:

* Pregnant or lactating women.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Modified Swiss Narcolepsy Scale total score < 0 at Screening or history of narcolepsy or cataplexy.
* Any contraindication to citalopram or any other selective serotonin reuptake inhibitor.
* History of cardiovascular disease (e.g., congenital long QT syndrome, arrhythmia).
* Relevant history of a suicide attempt or suicidal behavior.
* Personal or family history of psychiatric disorder(s).
* Individuals of Asian descent.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to Screening.
* Excessive caffeine consumption, defined as ≥ 800 mg per day at screening.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 2 weeks or 5 terminal half-lives (t½; whichever is longer) prior to first study treatment administration.
* Ongoing, recurrent, or chronic hypokalemia or hypomagnesemia.

Ages: 24 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline for Saccadic Peak Velocity (degrees/sec) to assess sedation | From pre-dose to 8 hours after dosing on Day 1, Day 2, Day 3, Day 9, and Day 10

OTHER OUTCOMES:
Number of participants with treatment-emergent AEs from study treatment administration up to EOS | AEs from Day 1 to EOS; for up to 15 days post-dose
Number of participants with treatment-emergent SAEs from study treatment administration up to EOS | SAEs from Day 1 to EOS; for up to 50 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Parexel International GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No